CLINICAL TRIAL: NCT05045729
Title: Incidence, Survival and EMS-treatment of Out-of-Hospital Cardiac Arrests Related to Exercise
Brief Title: OHCA Sports in Denmark
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: Region Sjælland (Other); Region Syddanmark (Other); Region MidtJylland Denmark (Other); North Denmark Region (Other Government); TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Helle Collatz, Associate professor, MD, PHD, Emergency Medical Services, Capital Region, Denmark
Other Study IDs: F-35101-01-SAWL
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Emergency Medical Services
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OHCA SPORTS: All OHCA, where the patient was engaged in sports at the time of the event

SUMMARY:
While regular exercise is known to prevent cardiovascular disorders, exercise might also trigger acute cardiac events such as cardiac arrest. This study examines the incidence, prognosis and outcomes of out-of-hospital cardiac arrest (OHCA) related to exercise in the general population of Denmark.

This retrospective cohort study examins all OHCAs in the Danish Cardiac Arrest Registry from 2016 to 2019 in Denmark. OHCA related to exercise were identified in the nationwide electronic database and coupled to the patient register. OHCA related to exercise was defined as occurring during or up to one hour after exercise of moderate or vigorous intensity. Descriptive statistics are used together with an adjusted multivariate logistic regression model to assess predefined factors of interest.

DETAILED DESCRIPTION:
The Danish Emergency Medical System (EMS) introduced a nationwide registry of electronic medical reports in 2016.(1) This report system allows electronic searches and thereby the opportunity to identify subgroups of out-of-hospital cardiac arrests (OHCA). Thus, this novel reporting enables the possibility to investigate new characteristics in OHCA related to exercise.

Exercise and physical activity have been shown to reduce the risk of cardiovascular disease, in spite of this, exercise can be related to a transient increased risk of cardiac events including sudden cardiac arrest.(2) Literature have reported low annual incidences of OHCA related to exercise between 0.48 - 2.1 per 100.000 person-years. (3-7) With the proportion of OHCA related to exercise of 0.3 - 7 % of all OHCA's (4,8,9). No standardized definition of timeframe concerning OHCA related to exercise is established, but throughout the literature onset of symptoms is defined to be during or up to one hour after exercise(4,5,10,11). Overall survival rates among previous studies varies from 11 - 46.2 % (6,12), a 30-day survival rate between 5.5 - 58 % (8,13) and a survival to discharge between 15.7 - 77 % (4,5,9,10,14). Yet, data is assessed in different countries with different health care systems, in different subgroups of age and lastly throughout different periods of time. This suggests further investigations and cohesion to standardized reporting, advocating for the Utstein Reporting Template. (15) Despite conflicting results regarding survival, there is consensus that exercise related OHCA has a better prognosis compared to OHCA not related to exercise. (4-6,8-10,16,17) Another consistent finding is younger age among patients suffering from OHCA related to exercise compared to other OHCA's. (5,6,9,10,17)

The etiology is often classified as either of (presumed) cardiac etiology or of non-cardiac etiology. (15) The Utstein Model suggests a method of which the pathogenesis is categorized under either medical (presumed cardiac or unknown or other medical i.e., gastro-intestinal bleed, anaphylaxis etc.) or traumatic cause, drug overdose, drowning, electrocution or asphyxia (external). If more than one cause is potential, the most likely should be noted.(18) In addition, it is suggested, that OHCA related to exercise often is caused by a presumed cardiac etiology. (4,5,7).

A better understanding and enhanced knowledge of the epidemiology of OHCA during exercise, could be useful for appropriate handling of these situations, thus this study aims to:

* Report the national incidence of exercise related OHCA's among cases attended by the Danish Medical Emergency System (EMS).
* To assess survival defined as return of spontaneous circulation (ROSC) and 30-day survival
* Finally, to evaluate aspects associated with better outcome including localization, observation of occurrence, bystander CPR, initial rhythm, use of defibrillator and patient demographics.

Materials and Methods This registry-based follow-up study includes data from patients in The Danish Medical Service electronical registry over a 4-year period from 2016-2019 with OHCA related to exercise.

Data Data on OHCA's with attempted resuscitation in Denmark have been collected in the electronic based Danish Medical Service reporting system since 2016. The registry covers detailed data including the EMS report. The data consists of executive entries and advanced text searches of prehospital charts in conjunction, augmenting the identification and collecting all OHCA's in Denmark. All cases have been through an elaborate validation process of which all identified events were read through manually. This was conducted by an external verification team to corroborate high quality of data throughout the approximately 5200 cases of OHCA in Denmark annually. Within this practice of verification, supplementary sources of data have been linked to each individual case of OHCA; information of certain interest was survival, localization, initiation of bystander CPR and actions from EMS personnel.

Identification of OHCA related to exercise This study evaluates OHCA related to exercise. All cases of OHCA were assessed and coupled to the electronic prehospital medical record, which, in context, facilitates advanced text searching in the complete electronic prehospital medical reporting system. Hence did the external validation team mark all charts consisting information about localization and type of exercise. All case descriptions in the prehospital medical records of OHCA occurring at sporting facilities were reviewed. Regarding events outside a sporting facility following terms were marked: Cases were categorized and afterwards classified in 6 subgroups; Team sports (Soccer, Handball, Volleyball, Tennis and Badminton), Fitness (Gymnastics, Aerobic, Cross Fit, Weight Lifting, Strength Training, Dancing, Yoga, Pilates, Athletics), Running/Jogging (Marathon, Ironman, Triathlon, Running, Jogging, Power walking, Roller-skating), Cycling (Cycling, Mountain Biking, Spinning), Water Sports (Swimming, Sailing, Surfing, Kitesurfing, Rowing, Kayaking) and lastly Miscellaneous (Bowling, Hunting, Golf, Equestrian sports) and their derivatives. (19,20) Furthermore time of onset of symptoms were marked in relation to the activity.

Identification of presumed causes Three individual raters will go through data to independently identify presumed causes of OHCA related to exercise. This evaluation will categorize cases as either presumed reversible or presumed non-reversible. Cases will be assessed based on the Utstein model regarding etiology. Including presumed cardiac or unknown or other medical, or traumatic cause, drug overdose, drowning, electrocution or asphyxia (external) etiology supported by a free-text description. Any discrepancy or ambiguity will be undertaken by third party members. Cases with lack of valuable information concerning cause or if several conflicting causalities is present will be labelled as "NA" or "Inconclusive" respectively. Contingent on an obviously causality between chronical disease and the presentation of the case and no plausible reversible causes, the case will be labelled non-reversible.

Variables included

* Age: Age will be defined as the subject age at the time of the event.
* Gender: Gender will be stated as either male, female or undetermined derived from personal identification numbers. Gender will be characterized based on EMS-charts, in those cases without an identification number.
* Initial rhythm: The initial rhythm will be defined as the first rhythm observed by EMS personnel, and categorized as either shockable, non-shockable (asystole), non-shockable (other) or undetermined.
* Etiology of cardiac arrest: Presumed causes will be stated as either presumed cardiac, other medical cause, trauma, drug overdose, drowning, electrocution or hypoxemia (external).
* Location of Incidence: Location will be characterized as either; sport facilities, gym, residential area, outdoors and nature, private home or other.
* Observation of occurrence: Cardiac arrests will be defined as either unwitnessed, bystander witnessed or EMS-witnessed.
* Cardio-pulmonary-resuscitation (CPR): CPR will include bystander-initiated CPR and EMS treatment with CPR.
* Defibrillation and use automatic external defibrillators (AEDs): Defibrillation will include defibrillation by bystanders and/or EMS personnel. Use of AED's includes using the device also in the case it did not deliver shocks.
* EMS-response time: This will be defined as the time between a dispatcher receiving the emergency call and the arrival of the first EMS-personnel.
* Hospitalization: Hospitalization will be considered as either; transported to hospital or declared dead by EMS-personnel.
* Return-of-spontaneous-circulation (ROSC): ROSC will be classified as the achievement of ROSC anytime between recognition of the event and termination (defined as either hospital admission or declaration of death by EMS-personnel).
* State at hospital admission: State of the case upon arrival at the hospital will be defined as either ROSC or ongoing CPR.
* Survival: Survival will be defined as ROSC at the time of hospital admission, additionally 30-day survival will be included, this derived from data from the National Patient Registry.

Analysis All data will be pseudo-anonymized, and all analyses will be accomplished on an aggregated nationwide level. Data is collected using the STrengthening the Reporting of OBservational studies in Epidemiology (STROBE) statement. The objective of this study is to clarify etiology, descriptive data and prehospital interventions of OHCA's related to exercise. Secondary an update of the annual incidence and survival rate is carried out. Descriptive statistics includes the above-mentioned variables labelled with absolute numbers and percentages. Comparative analyses will be carried out using non-parametric testing to examine subgroups. Forward logistic regression analysis will be performed for multivariate analysis. Odds ratio for survival will be calculated stratified by etiology, localization, bystander and EMS-actions.

Data storage Data is stored on secure drive according to the regional instructions for safe conduct of data management.

Ethical considerations GDPR will be followed according to danish law and the study is registered and approved at the Danish Data Protection Agency, capital region of Denmark (reference 2007-58-0015, GEH-2014-019, I-suite 02737). Since it is a registry-based study, no ethical approval is required.

Perspectives This study provides novel information regarding OHCA related to exercise; the descriptive statistics provides relevant data based on a reviewed, high-quality database. Furthermore, throughout analyses, a better understanding of the preceding circumstances and etiology might contribute to improve handling this type of arrests. This, eventually through the use of campaigns targeted laypersons and healthcare personnel.

Publication The final results are targeted for publication in an international peer reviewed journal. Participation as coauthors will be decided according to the Vancouver criteria or acknowledged for providing access to data. All Danish regional EMS regions will receive this manuscript prior to publication for eventual comments.

List of Abbreviations AED: Automatic External Defibrillator CPR: Cardio Pulmonary Resuscitation EMS: Emergency Medical Services GDPR: General Data Protection Regulation OHCA: Out-of-Hospital Cardiac Arrest ROSC: Return of Spontanous Circulation STROBE: STrengthening the Reporting of OBservational studies in Epidemiology

References

1. Lindskou TA, Mikkelsen S, Christensen EF, Hansen PA, Jørgensen G, Hendriksen OM, et al. The Danish prehospital emergency healthcare system and research possibilities. Scand J trauma, Resusc Emerg Med. 2019;27(1):100.
2. Friedewald VE, Spence DW. Sudden cardiac death associated with exercise: the risk-benefit issue. Am J Cardiol. 1990;66(2):183-8.
3. Marijon E, Bougouin W, Celermajer DS, Perier M-C, Benameur N, Lamhaut L, et al. Major regional disparities in outcomes after sudden cardiac arrest during sports. Eur Hear journal. 2013;34(47):3632-40.
4. Eastwood D, Andrew E, Smith K, Nair R, Nehme Z, Bernard S, et al. Exercise-related out-of-hospital cardiac arrest in Victoria, Australia. Resuscitation. 2019;139:57-64.
5. Edwards MJ, Fothergill RT. Exercise-related sudden cardiac arrest in London: incidence, survival and bystander response. Open Hear. 2(1):e000281.
6. Berdowski J, de Beus MF, Blom M, Bardai A, Bots ML, Doevendans PA, et al. Exercise-related out-of-hospital cardiac arrest in the general population: incidence and prognosis. Eur Hear journal. 2013;34(47):3616-23.
7. Holst AG, Winkel BG, Theilade J, Kristensen IB, Thomsen JL, Ottesen GL, et al. Incidence and etiology of sports-related sudden cardiac death in Denmark-Implications for preparticipation screening. Hear Rhythm. 2010 Oct;7(10).
8. Kiyohara K, Sado J, Matsuyama T, Nishiyama C, Kobayashi D, Kiguchi T, et al. Out-of-hospital cardiac arrests during exercise among urban inhabitants in Japan: Insights from a population-based registry of Osaka City. Resuscitation. 2017;117:14-7.
9. Søholm H, Kjaergaard J, Thomsen JH, Bro-Jeppesen J, Lippert FK, Køber L, et al. Myocardial infarction is a frequent cause of exercise-related resuscitated out-of-hospital cardiac arrest in a general non-athletic population. Resuscitation. 85(11):1612-8.
10. Toukola TM, Kauppila JP, Pakanen L, Kortelainen M-L, Martikainen M, Huikuri H V., et al. Characteristics and Prognosis of Exercise-Related Sudden Cardiac Arrest. Front Cardiovasc Med. 2018 Jul 26;5.
11. Rai M, Thompson PD. The definition of exertion-related cardiac events. Br J Sports Med. 2011 Feb 1;45(2).
12. Drezner JA, Chun JSDY, Harmon KG, Derminer L. Survival trends in the United States following exercise-related sudden cardiac arrest in the youth: 2000-2006. Hear Rhythm. 5(6):794-9.
13. Si Oon Cheah, Marcus E H Ong MBFC. An eight year review of exercise-related cardiac arrests. Ann Acad Med Singap. 2010;
14. Marijon E, Tafflet M, Celermajer DS, Dumas F, Perier M-C, Mustafic H, et al. Sports-Related Sudden Death in the General Population. Circulation. 2011 Aug 9;124(6).
15. Cummins RO, Chamberlain DA, Abramson NS, Allen M, Baskett PJ, Becker L, et al. Recommended guidelines for uniform reporting of data from out-of-hospital cardiac arrest: the Utstein Style. A statement for health professionals from a task force of the American Heart Association, the European Resuscitation Council, the Heart and Stroke Foundation of Canada, and the Australian Resuscitation Council. Circulation. 1991 Aug;84(2).
16. Marijon E, Uy-Evanado A, Reinier K, Teodorescu C, Narayanan K, Jouven X, et al. Sudden cardiac arrest during sports activity in middle age. Circ J Am Hear Assoc. 131(16):1384-91.
17. Page RL, Husain S, White LY, Rea TD, Fahrenbruch C, Yin L, et al. Cardiac arrest at exercise facilities: implications for placement of automated external defibrillators. J Am Coll Cardiol. 62(22):2102-9.
18. Perkins GD, Jacobs IG, Nadkarni VM, Berg RA, Bhanji F, Biarent D, et al. Cardiac Arrest and Cardiopulmonary Resuscitation Outcome Reports: Update of the Utstein Resuscitation Registry Templates for Out-of-Hospital Cardiac Arrest. Circulation. 2015 Sep 29;132(13).
19. Danmarks statistik. https://www.statistikbanken.dk/10673.
20. Idrættens Analyseinstitut. https://www.idan.dk/vidensbank/downloads/danskernes-motions-og-sportsvaner-2016/9a94e44b-4cf5-4fbe-ac89-a696011583d5. 2016.

ELIGIBILITY:
Inclusion Criteria:

* OHCA

Exclusion Criteria:

* EMS witnessed OHCA

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This registry-based follow-up study includes data from patients in The Danish Medical Service electronical registry over a 4-year period from 2016-2019 with OHCA related to exercise.
Sampling Method: Non-Probability Sample
Enrollment: 21298 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 30 days
  Patients survival after OHCA

SECONDARY OUTCOMES:
ROSC | Prior to hospital admittance
  Patient obtains return of spontaneous circulation

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request